CLINICAL TRIAL: NCT06494085
Title: PressUre-Muscle-index to Identify Patient's Desired Tidal Volume and the Threshold of Over-Assistance During Pressure Support Ventilation
Brief Title: Pressure Muscle Index and Threshold of Over-assistance During Pressure Support Ventilation
Acronym: PUMA
Status: Recruiting | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 24-105
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2024-08

CONDITIONS: Acute Hypoxemic Respiratory Failure
Keywords: Mechanical Ventilation; Intensive Care Unit; Pendelluft; Pressure Support Ventilation
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Measuring Respiratory Mechanics — First, for each patient enrolled we will perform inspiratory and expiratory occlusions - routinely performed diagnostic maneuvers to measure patient's breathing effort - at the clinically set level of breathing assistance by the mechanical ventilator. Importantly, we will measure pressure-muscle-index (PMI).
  Second, we will set the level of assistance (i.e. pressure support, PS) in order to make PMI=0. The PS level at which PMI=0 (PS PMI=0) will be used as reference for the study protocol. After 5 minutes at PS PMI=0 we will perform inspiratory and expiratory occlusions.
Other: Randomized Pressure Support — 3 steps of PS above (+2, +4, +6 cmH2O) and 3 below (-2, -4, -6 cmH2O) PSPMI=0 done in a randomized order (sequence in envelopes opened blindly by the investigators). Each step will last ≤5 minutes if poorly tolerated (see tolerance rule in description). At the end of each step we will perform 1 inspiratory occlusion and 3 expiratory occlusions. Each of the expiratory occlusion will be separated by 30 seconds in order to restore the patient's breathing pattern. We will resume a 3-minutes clinical PS in between each step to minimize changes in PaCO2. If not yet comprised by the study steps each patient will undergo an adjunctive 5 minutes step at PS 0 (zero) cmH2O.

SUMMARY:
Pressure support ventilation (PSV) is used to assist the breathing of the intubated patient with some pressure from the ventilator. This support aims at avoiding excessive inspiratory effort, while ensuring a certain degree of training of the patient's inspiratory muscle. Avoiding both minimal and excessive assistance is thus important for the optimal care of the intubated patient ensuring a lung and diaphragm protective ventilation with the goal to liberate the patient from the ventilator as soon as possible.

Recently pressure-muscle-index (PMI), an index of inspiratory effort easy to be measured on the ventilator screen, has been proposed to avoid excessive assistance in PSV. This will be the first prospective study testing the effects of setting pressure support based on PMI to avoid excessive assistance on patients recovering from acute lung injury (acute hypoxemic respiratory failure).

DETAILED DESCRIPTION:
First, for each patient enrolled the investigators will perform 1 inspiratory and 3 expiratory occlusions separated at least by 30 seconds at clinical PSV to measure respiratory mechanics (plateau pressure [Pplat] and respiratory system compliance [Crs] and elastance [Ers]) and inspiratory effort and drive (Pocc, P0.1, PMI) and Vt expressed in ml/Kg of predicted body weight.

Second, if PMI≥0 at baseline, the investigators will set Pressure Support (PS) so that positive end-expiratory pressure (PEEP) +PS (i.e. Peak pressure [Ppeak]) equals Pplat measured at baseline, in order to make PMI=0. If PMI<0 at baseline, the investigators will set PS so that PEEP+PS equals Pplat measured at baseline, then the investigators will perform an inspiratory occlusion and repeat the procedure until PMI=0. The PS level at which PMI=0 (PSPMI=0) and the corresponding breathing pattern (tial volume [Vt] and respiratory rate [RR]) will be used as reference for the study protocol. After 5 minutes at PSPMI=0 the investigators will perform 3 inspiratory and 3 expiratory occlusions separated at least by 30 seconds.

Third, each patient will undergo 3 steps of PS above (+2, +4, +6 cmH2O) and 3 below (-2, -4, -6 cmH2O) PSPMI=0 in a randomized order. Steps will be randomized using a simple sequence written within envelopes opened blindly by the investigators. Each step will last 5 minutes or less if poorly tolerated (see tolerance rules below). At the end of each step the investigators will perform 1 inspiratory occlusion and 3 expiratory occlusions. Each of the expiratory occlusion will be separated by 30 seconds in order to restore the patient's breathing pattern. The investigators will resume a 3-minutes clinical PS in between each step to minimize changes in PaCO2. If not yet comprised by the study steps each patient will undergo an adjunctive 5 minutes step at PS 0 (zero) cmH2O.

The study protocol will last approximately 60 minutes. The patient will be continuously monitored by a physician and a respiratory therapist.

At the end of the study, if different from clinically set PS, the investigators will propose clinicians to adjust the PS to target PMI>0 and a lung and diaphragm protective ventilation strategy following current literature. Data about PS setting at the end of the study will be recorded in the case report form.

Tolerance rules:

Protocol will be stopped if: heart rate >140 beats/min; increase in respiratory rate by 50% or more if not explained by ineffective effort; hypotension [systolic blood pressure <90 mmHg] or hypertension [systolic blood pressure >180 mmHg]; peripheral arterial oxygen saturation <90% for 5 minutes; excessive use of accessory respiratory muscles, diaphoresis, agitation, and the appearance of major abdominal or thoracic paradoxical movements. If apnea would appear at high PS levels (as described as overassistance), the PS will be decreased to the next lower level. PS will be set to not exceed a Ppeak of 30 cmH2O or a Vt of 12 mL/kg of predicted bodyweight

ELIGIBILITY:
Inclusion Criteria:

* >18 y.o.
* Invasively ventilated in Intensive Care Unit.
* Diagnosed with acute hypoxemic respiratory failure (P/F<300 mmHg).
* Breathing on pressure support ventilation.

Exclusion Criteria:

* <18 y.o.
* Contraindication for Electrical Impedence Tomography monitoring (e.g. pacemaker, burns, or - wounds limiting electrode placement).
* Severe and previously diagnosed neurological and neuromuscular disease.
* Psychomotor agitation (Sedation Agitation Scale > 4).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Study population will include patients mechanically ventilated in the St. Michael's Intensive Care Unit. Patients who are younger than 18 years of age will be excluded from this study on the basis that the ICUs at St. Michael's Hospital are intended for adults; individuals aged less than 18 years are rarely, if ever, admitted.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Inspiratory Occlusion | 60 minutes
  To investigate the role of the inspiratory occlusion as a diagnostic tool to understand the patient's desired tidal volume and minute ventilation in Pressure Support Ventilation (PSV),
Pressure Muscle Index (PMI) | 60 minutes
  To investigate the role of a PMI>0 strategy to avoid over-assistance in Pressure Support Ventilation

SECONDARY OUTCOMES:
Pendelluft | 60 minutes
  To investigate the relationship between "active" and "passive" pendelluft measured over different levels of assistance in PSV.
Lung and Diaphragm Protective Ventilation | 60 minutes
  To measure indexes proposed by current literature to target a lung and diaphragm protective ventilation strategy with both inspiratory and expiratory occlusions in PSV, while applying a PMI>0 strategy.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Brochard, Principal Investigator — Unity Health Toronto - St. Michael's Hospital
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No